CLINICAL TRIAL: NCT04423042
Title: A Nested Interventional Cohort Study to Assess the Efficacy and Safety of Adjunctive Humanized Monoclonal Interleukin-6 Receptor Blocker Tocilizumab (TCZ) Therapy to Standard of Care for the Reduction of Hyperinflammation Related Mortality in SARS-Cov2 Positive Patients
Brief Title: Tocilizumab in Coronavirus-19 Positive Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0713
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Covid19; COVID-19; Severe Acute Respiratory Syndrome Coronavirus 2; Coronavirus; Inflammation
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Inflammation | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab Arm (Experimental): Tocilizumab 8 mg/kg IV up to a maximum of 800 mg with possible repetition of the same dosage within 28 hours (the optional second dose after 12 hours but before 28 hours following the first dose), based on the clinical judgement of the attending physician in consultation with the COVID-inflammation team.
  Interventions: Biological: Tocilizumab
- No Intervention Arm (No Intervention): No intervention arm patients will be identified from medical records, as being COVID-19 positive patients with hyperinflammation who did not receive any interleukin antagonist treatment.

INTERVENTIONS:
Biological: Tocilizumab — Tocilizumab binds to both soluble and membrane-bound interleukin-6 receptors and has been shown to inhibit interleukin 6-mediated signalling.
  Other Names: Actemra
  Arms: Tocilizumab Arm

SUMMARY:
This is a cohort study of COVID-19 patients with hyperinflammation. It aims to determine the impact of adjunctive Tocilizumab (TCZ) to standard of care on the reduction of hyperinflammation-related mortality in COVID-19. Patients with COVID-19 are at high risk of life-threatening hyperinflammation and death. One in three COVID-19 patients admitted to ICU was found to develop life-threatening hyperinflammation. The risk of death when untreated is estimated to be 50-80%.

DETAILED DESCRIPTION:
The novel coronavirus, SARS-Cov2/COVID-19, emerged in late 2019 in Wuhan, China. Quickly, SARS-CoV2 spread to all corners of the globe. In March 2020, The World Health Organization (WHO) declared SARS-CoV2/COVID-19 a pandemic. Individuals infected with SARS-CoV2 have a varied clinical presentation, ranging from asymptomatic or mild respiratory symptoms to severe involvement of the lower respiratory tract, with patients requiring mechanical ventilation. A particular point of interest is how the overall severity and clinical outcomes of COVID-19 patients may be associated with the excessive production of pro-inflammatory cytokines, or hyperinflammation, leading to acute respiratory distress syndrome. This state of hyperinflammation may be associated with increased mortality in COVID-19 patients. Tocilizumab, an Interleukin-6 antagonist, may help treat COVID-19 associated hyperinflammation.

This is a nested interventional cohort study of COVID-19 patients with hyperinflammation. It aims to determine the impact of adjunctive Tocilizumab (TCZ) to standard of care on the reduction of hyperinflammation-related mortality in COVID-19. Patients with COVID-19 are at high risk of life-threatening hyperinflammation and death. One in three COVID-19 patients admitted to ICU was found to develop life-threatening hyperinflammation. The risk of death when untreated is estimated to be 50-80%. TCZ treatment may reduce mortality.

Primary objective: To establish that tocilizumab, in addition to standard of care, reduces the 30-day mortality from hyperinflammation in COVID-19 disease significantly compared to no anti-interleukin therapy plus standard of care.

Secondary objectives: To evaluate the addition of tocilizumab therapy to standard of care on a number of secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. All genders
3. Hospitalization for suspected or confirmed SARS-CoV2 infection. COVID-19 diagnosis defined as positive on reverse-transcriptase polymerase chain reaction, with provincial laboratory confirmation.
4. Signs of hyperinflammation (cytokine release syndrome) defined by the presence of any of the following:

   i. Elevated C-reactive protein (≥70 mg/dl and/or rising since last 24h not due to bacterial infection), ii. Ferritin (>700 mcg/L and/or rising since last 24h),
5. Anti-interleukin treatment indication as per hyperinflammation team
6. Informed consent for participation in the study

Exclusion Criteria:

1. Goal of Care C (palliative care)
2. Known hypersensitivity to TCZ or its components
3. Current systemic immunosuppressive therapy; anti-interleukin 1 or anti-interleukin 6 treatment
4. Known active bacterial or fungal infections or other clinical conditions that contraindicate TCZ and cannot be treated or resolved according to the physician's judgment
5. Current or history of bowel perforation or diverticulitis
6. Suspicion of active or latent tuberculosis
7. Pregnant or breastfeeding patient
8. Patients with known prior liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-30 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Assessed at 30 days post treatment
  Mortality status of participants

SECONDARY OUTCOMES:
Ordinal Scale for evaluating subject clinical status at days 3, 8, 15, 30, 60 post treatment. | Assessed at days 3, 8, 15, 30, 60 post treatment
  Uninfected, ambulatory, hospitalized: mild disease, hospitalized: severe disease, death

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Benseler, MD PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
Results will be rapidly published.

REFERENCES:
- [Background] Xu X, Han M, Li T, Sun W, Wang D, Fu B, Zhou Y, Zheng X, Yang Y, Li X, Zhang X, Pan A, Wei H. Effective treatment of severe COVID-19 patients with tocilizumab. Proc Natl Acad Sci U S A. 2020 May 19;117(20):10970-10975. doi: 10.1073/pnas.2005615117. Epub 2020 Apr 29. PMID 32350134
- [Background] Alzghari SK, Acuna VS. Supportive Treatment with Tocilizumab for COVID-19: A Systematic Review. J Clin Virol. 2020 Jun;127:104380. doi: 10.1016/j.jcv.2020.104380. Epub 2020 Apr 21. No abstract available. PMID 32353761
- [Background] Zhang C, Wu Z, Li JW, Zhao H, Wang GQ. Cytokine release syndrome in severe COVID-19: interleukin-6 receptor antagonist tocilizumab may be the key to reduce mortality. Int J Antimicrob Agents. 2020 May;55(5):105954. doi: 10.1016/j.ijantimicag.2020.105954. Epub 2020 Mar 29. PMID 32234467
- See also: Hoffmann-La Roche Limited. Product Monograph, ACTEMRA® tocilizumab. — https://www.rochecanada.com/PMs/Actemra/Actemra_PM_E.pdf